CLINICAL TRIAL: NCT02907697
Title: Adherence Intervention for HIV-infected Drug Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Kasey Claborn, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23DA039037 (NIH)
Record Dates: First submitted 2016-08-26; First posted 2016-09-20 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: HIV; Substance Use
Keywords: HIV/AIDS; adherence; substance use; HIV care continuum
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LifeSteps-Drug Use (Experimental): The investigators expect the LifeSteps-Drug Use adaptation will be modeled after the Life Steps adherence intervention with the addition of a Drug Use module based on motivational interviewing and the FRAMES approach. The LifeSteps-Drug Use intervention is expected to include two in-person sessions and two telephone booster sessions. While anticipated preliminary adaptations have been based on the extant literature, changes to the protocol will be based on data obtained during the qualitative phase which will be sufficiently broad and open to assess for factors that we have not anticipated.
  Interventions: Behavioral: Life Steps-Drug Use
- Health Education (Active Comparator): The health education condition is a time-matched, active control arm. It will consist of two in-person sessions and two telephone sessions. Each session will cover a general health education topic.
  Interventions: Behavioral: General Health Education

INTERVENTIONS:
Behavioral: Life Steps-Drug Use
  Arms: LifeSteps-Drug Use
Behavioral: General Health Education
  Arms: Health Education

SUMMARY:
Many people living with HIV use illicit drugs, which leads to worsened health outcomes and increased transmission of HIV due to poor adherence to medication regimens. This research will develop an intervention targeting medication adherence that is tailored to the unique needs of HIV-infected drug users. This research will promote adherence and improve treatment outcomes among HIV-infected drug users thereby minimizing the development of drug resistant strains of HIV and reducing transmission.

DETAILED DESCRIPTION:
This K23 research and training award advances the long-term goal of improving treatment outcomes and reducing transmission of HIV among HIV-infected drug users. The proposed training and research plans will enable the PI to develop the skills needed for an independent research career in the area of illicit drug use and HIV adherence intervention. The objective of this award is to develop skills in implementation science, behavioral intervention development and evaluation with drug using populations, and in-depth qualitative data analysis to accelerate refinement and effective implementation of interventions for HIV-infected drug users. Multiple comorbidities such as drug use and HIV act synergistically to produce poorer health outcomes and increase morbidity, mortality, and transmission of HIV. Consequently, effective and sustainable interventions adapted to drug users to improve antiretroviral medication adherence and reduce risk behaviors are urgently needed. Drug users present unique treatment challenges compared with other HIV-infected populations, including lower rates of adherence and inferior treatment outcomes. Additionally, interpersonal factors, including social support, negative patient-provider interactions, and socioeconomic challenges present significant barriers to adherence. Thus, the generalizability of current adherence interventions to drug users is limited, and there is a pressing need for efficacious interventions adapted to HIV-infected drug using populations. This project addresses this gap by being the first to adapt and test the acceptability and efficacy of a combined adherence and brief motivational intervention for HIV-infected drug users. Specifically, the intervention will augment the established Life Steps adherence intervention to include: (1) a tailored Life Steps module addressing the unique needs of illicit drug users, aimed at improving medication adherence; (2) a brief Motivational Interview to address drug use and other risk behaviors; and (3) two follow-up booster sessions. A three-phase, top-down research approach to adapt, refine, and pilot test the intervention will be conducted. Phase 1 will include focus groups with HIV-infected drug users currently prescribed antiretroviral medications and individual interviews with community-based clinicians. Phase 2 will include manual development, therapist training, a pilot trial, in-depth qualitative interviews, and further manual revisions. Phase 3 will include a small, 2-armed (intervention vs. health education control) randomized controlled trial with 60 HIV-infected drug users. Feasibility, acceptability, and preliminary indication of improvement in antiretroviral adherence and reduction in drug use will be examined at 1-, 3-, and 6-month follow-ups. To enable the PI to pursue this long-term research agenda, she will work with experienced mentors to build three areas of expertise: (1) proficiency in qualitative research methods and analysis; (2) skills in intervention development and evaluation with illicit drug using populations; (3) expertise in advanced longitudinal data analysis; and (4) implementation science. This K23 study addresses a key priority in HIV treatment science, and it will fully prepare the PI for an independent research career as an HIV intervention scientist.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* HIV-infected
* prescribed an antiretroviral regimen
* meet DSM-V criteria for a substance use disorder (other than tobacco and alcohol) and report ≥3 days of use of an illicit drug per month over the past 90 days.
* self-report <100% adherence and have experienced a detectable viral load (>20 copies/mL) within the last 6 months.

Exclusion Criteria:

* cognitive impairments that jeopardize informed consent
* active psychosis
* current suicidal ideation
* not fluent in English
* have a prescription for and report only medicinal use of marijuana

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Antiretroviral Adherence | 1-, 3-, and 6-months
  Change in Antiretroviral Adherence will be assessed by use of medical event monitoring systems (MEMS). MEMS is a pill-bottle-cap with a pressure activated chip which records time/date the bottle is opened. MEMS data will be collected on one antiretroviral medication following a triage criterion established in studies of antiretroviral adherence.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D) | 1-, 3-, and 6-months
  Change in depression over time will be assessed using the Center for Epidemiologic Studies Depression Scale (CES-D) is a widely used 20-item measure and has good sensitivity and specificity and high internal consistency and has been used extensively with PLWH and is related to ART adherence.
HIV Treatment Adherence Self-Efficacy (HIV-ASES) | 1-, 3-, and 6-months
  Change in treatment self-efficacy will be assessed using the HIV-ASES whic is a 12-item scale of patient confidence in their ability to carry out behaviors related to adhering to medication regimens.
U.S. Health Resources and Service Administration measure of HIV treatment retention | 1-, 6-months
  Change in HIV Treatment Retention will be measured with the U.S. Health Resources and Service Administration measure of HIV treatment retention, which defines treatment retention as having at least two outpatient visits separated by at least 90 days during a 12-month period
Risk Assessment Battery | 1-, 3-, and 6-months
  Change in HIV risk behavior will be assessed using the Risk Assessment Battery which assesses HIV risk behavior, including sex risk and drug risk, in the past six months.
HIV1 Ultra RT PCR-Roche test | 1-, 3-, and 6-months
  This lab assay will be used to assess change in HIV viral load over time.
Urine Toxicology Screens | 1-, 3-, and 6-months
  Participants will be asked to give a urine sample at each assessment. Redwood Toxicology Redi-cups urine drug screens have test strips in the specimen lids allowing for fast screening without spillage. The Redi-cups 5-panel urine drug screen tests for cocaine, THC, methamphetamines, opiates, and benzodiazepines. This will provide biological verification of drug use to assess change in drug use over time.
ACTG Self-Reported Antiretroviral Medication Adherence | 1-, 3-, and 6-months
  The ACTG scale will be used to assess self-reported adherence to antiretroviral medications.
30-day Timeline Followback (TLFB) | 1-, 3-, and 6-months
  The TLFB will be used to assess change in alcohol, tobacco, and illicit drugs over time.

CONTACTS AND LOCATIONS:
Overall Officials: Kasey Claborn, PhD, Principal Investigator — The Unviersity of Texas
Locations (1):
- Unviersity of Texas Dell Medical School, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Claborn K, Becker S, Operario D, Safren S, Rich JD, Ramsey S. Adherence intervention for HIV-infected persons who use drugs: adaptation, open trial, and pilot randomized hybrid type 1 trial protocol. Addict Sci Clin Pract. 2018 Apr 2;13(1):12. doi: 10.1186/s13722-018-0113-5. PMID 29606129